CLINICAL TRIAL: NCT07200518
Title: The Multistrain Probiotic OMNi-BiOTiC® Hetox for Treatment After Neurosurgery (ProSURG)
Brief Title: Effect of Probiotics After Neurosurgery
Acronym: ProSURG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Maribor (Other)
Collaborators: University Medical Centre Maribor (Other)
Responsible Party: Principal Investigator, Sabina Fijan, Full prof. dr., University Maribor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UKC-MB-KME-38/24
Record Dates: First submitted 2025-09-18; First posted 2025-10-01 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Healing
Keywords: neurosurgery; probiotics; Omni-Biotic Hetox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Lacticaseibacillus casei W56 Lactobacillus acidophilus W37 Levilactobacillus brevis W63 Lactococcus lactis W58 Lactococcus lactis W19 Bifidobacterium lactis W52 Ligiactobacillus salivarius W24 Bifidobacterium lactis W51 Bifidobacterium bifidum W23 corn starch, maltodextrin, plant protein, potassium chloride, magnesium sulphate, amylase manganese sulphate
  Interventions: Dietary Supplement: OMNi-BiOTiC® Hetox multistrain probiotic
- Placebo (Placebo Comparator): corn starch, maltodextrin, plant protein, potassium chloride, magnesium sulphate, amylase manganese sulphate
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: OMNi-BiOTiC® Hetox multistrain probiotic — OMNi-BiOTiC® Hetox multistrain probiotic
  Arms: Probiotic
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The goal of this randomised controlled trial is to determine the effect of consuming a multistrain probiotic OMNi-BiOTiC® Hetox on improving the healing, pain management, and postsurgical complications after neurosurgery.

The main question it aims to answer is:

• Is the multistrain probiotic OMNi-BiOTiC® Hetox effective in in improving patient-reported disability after neurosurgery?

Researchers will compare the probiotic group and the placebo group to determine if the healing is significantly different between the groups.

ELIGIBILITY:
Inclusion Criteria:

* adults with MRI-confirmed disc herniation, stenosis, or instability of the lumbar or cervical spine.
* Able to provide written informed consent
* Willing to comply with study procedures and follow-up assessments
* No contraindications to probiotic administration

Exclusion Criteria:

* symptoms of acute infection (vomiting, fever above 38°C, diarrhea, respiratory symptoms),
* chronic diseases,
* use of probiotics one month before inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Oswestry Disability Index (ODI) at 3 months | 4 weeks supplementation
  Functional disability will be assessed using the Oswestry Disability Index (ODI, version 2.1a; range 0-100, higher = greater disability). The primary outcome is the mean change in ODI from baseline to 3 months post-neurosurgery.

CONTACTS AND LOCATIONS:
Overall Officials: TOMAŽ ŠMIGOC, dr. med., Study Director — University Medical Centre Maribor; Sabina Fijan, Ph.D., Study Director — University of Maribor
Locations (1):
- University Medical Centre Maribor, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided